CLINICAL TRIAL: NCT00593398
Title: Malarial Immunity in Pregnant Cameroonian Women
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Diane Wallace Taylor, Professor, University of Hawaii
Other Study IDs: 07-0010
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria; pregnant women; infants; Cameroon
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples and biopsies of placental tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Malaria is caused by a parasite and is a health problem for mothers and fetuses (unborn infants). The Cameroonian Ministry of Health recommends that all pregnant women should take the drug sulfadoxine-pyrimethamine (also known as SP) every two months during pregnancy to avoid malaria. The purpose of this study is to find out how effective SP is in preventing pregnant Cameroonian women from getting malaria. Additional goals of this study are to see whether: SP prevents malaria parasites from causing changes in the placenta; SP prevents or helps women make a substance that keeps parasites from accumulating in the placenta; and whether SP affects the amount of protection a mother transfers to her baby. Participants will include 1,160 pregnant women, ages 15-50 years, and 216 babies born residing in Ngalii II and Ntouessong. Study procedures will include monthly blood samples from pregnant women and babies. Volunteers may participate in this study for up to 19 months.

DETAILED DESCRIPTION:
Plasmodium falciparum malaria is one of the three major infectious diseases in the world today. Infants in endemic areas are born with transplacentally-acquired antibodies (Ab) that help to protect them against severe infections. Once this passive-immunity wanes, infants become susceptible to severe disease. Asymptomatic and clinical malaria are more common in pregnant women, creating a health problem for both mother and developing fetus. Malaria increases maternal anemia, mortality at parturition and the risk of having low birth weight (LBW) babies. This study plans to enroll a total of 1,160 pregnant women, ages 15 to 50 years, including 920 pregnant women who reside in the city of Yaounde and 240 women who reside in the rural villages of Ngali II and Ntouessong. In addition, 216 babies born residing in Ngali II and Ntouessong will be enrolled. Women will receive physical exams, participate in blood sample collection, and will be followed monthly through their pregnancy. Participants will receive sulfadoxine - pyrimethamine (SP) every other month until term, as recommended by the World Health Organization (WHO). During the 2nd or 3rd visit, pregnant women will be asked to provide a stool sample for detection of intestinal parasites. At delivery, the following will be collected: 2-3 cc of maternal venous blood, information on the newborn, a biopsy of the placenta for histology, blood from the intervillous space of the placenta (IVS) for cytokines, and fetal cord blood for Ab and primed T and B cells. To determine how malarial infection during the 2nd and 3rd trimesters influences malarial infection in infants, mothers in the above study as well as additional mothers who received Intermittent Preventive Therapy (IPT)-SP during the 2nd and 3rd trimester and women who received less than the recommended dose will be recruited during their last trimester of pregnancy and asked to enroll their newborns. The levels of antimalarial cellular and humoral immunity at birth will be recorded for each infant. The newborn will be followed to determine when they 1st become positive for P. falciparum and the number and severity of infections. In addition, the decline of maternal Ab and acquisition of Ab (IgM and IgG) by infants to vaccine-candidate antigen (Ag) will be monitored throughout the 1st year using blood samples collected monthly. The goals of this study are to determine if the absence of malaria during the 2nd and 3rd trimesters (due to the use of IPT) does the following: alters the development of pregnancy-associated immunity in the mother; reduces placental pathology; and increases the susceptibility of babies to malaria. The primary outcome measures will be to determine: at delivery, the proportion of primigravidae with Ab to variant antigen identified by Salanti (VAR2csa) will be significantly reduced if pregnant women are not infected during the 3rd trimester of pregnancy; prevalence of presence of severe pathology will be compared among the groups; and the number of babies who have malaria during the first 6 months of life. The secondary outcome measures of this study will include: determining if maternal P. falciparum infection during the 2nd or 3rd trimester reduces the transfer of malaria-specific IgG to the fetus; determining if the proportion of babies who are born with primed T cells is the same in those whose mothers had malaria during the 2nd or 3rd trimester compared to those who did not; presence of primed B cells in cord blood will be detected by culturing cord blood mononuclear cells MNC in vitro culture for 5 days; and plasma collected from babies when they experience their 1st P. falciparum infection will be screened for the presence of IgG and IgM Abs against the panel of Ag. The duration of the entire study is 5 years.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who will be followed longitudinally during pregnancy:

* Greater than or equal to 15 years of age.
* Willingness to provide informed consent.
* Confirmed pregnancy.
* All gestational ages. Women less than 16 weeks of pregnancy will be enrolled, but they will not receive intermittent preventive therapy using sulfadoxine plus pyrimethamine (IPT-SP) until the 16th week of pregnancy or thereafter.
* Long-term residence in Yaounde, Ngali II or Ntouessong.
* Willingness of a women residing in Yaounde to release HIV testing results, obtained through a service provided by the MOH, to Dr. Leke, Cam-PI.
* Women residing in Ngalii II and Ntouessong will be encouraged to be HIV tested and asked to provide data on their HIV status to the project. However, HIV testing and providing the results will be optional.

Pregnant women enrolled near term:

* Same as above.
* Women who have a health booklet with entries entered by a physician/midwife/pharmacist about antimalarial treatment they have received during pregnancy

Inclusion criteria for infants living in Ngali II and Ntouessong:

* Resident of Ngali II or Ntouessong.
* Willingness of the mother/caregivers to give informed consent for their babies.
* Agree to bring the baby to the clinic whenever s/he becomes ill. Alternatively, inform the designated staff member or village health care worker that the baby is ill.
* Willingness to bring the baby for all recommended routine child-hood immunizations.
* Agree to provide a stool sample from the baby when s/he is 6 and 12 months of age.
* Twins will be included in the study.

Exclusion Criteria:

Pregnant Cameroonian women following longitudinally during pregnancy:

* Women who report a history of allergic reactions to sulfamides
* Women who report reactions to previously unknown antimalarial drugs
* Women with serious liver attacks (e.g., chronic hepatitis) or kidney failure or neurological conditions (e.g., seizures).
* Women with history of skin allergies
* Other conditions that in the opinion of the Director of Clinical Studies (DCS) or clinical staff (CS) would jeopardize the safety and rights of a participant in the trial or would render the participant unable to comply with the protocol.

Pregnant women enrolled near term:

* None.

Infants living in Ngali II and Ntouessong:

* Vague or incomplete information on maternal use of anti-malarials during pregnancy.
* Failure to inform the project staff that they are about to, or have delivered their babies, thereby preventing access to baseline information and specimens at birth that are critical for conduct of the study.
* Other conditions that in the opinion of the DCS, CS, or Cam-PI would jeopardize the safety and rights of a participant in the trial or would render the participant unable to comply with the protocol.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cameroonian women who are pregnant and living in the city of Yaounde or the village of Ngali II and Ntouessong in Soa district
Sampling Method: Non-Probability Sample
Enrollment: 990 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane W Taylor, PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Yaounde 1, Yaoundé, Cameroon